CLINICAL TRIAL: NCT03222869
Title: Assessment of Primary Oxygenation and Airflow Measurement for Endoscopic Laryngeal Surgery
Status: Completed | Type: Observational
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Other Study IDs: IRB00096150
Record Dates: First submitted 2017-07-18; First posted 2017-07-19 (Actual); Last update posted 2023-10-13 (Actual); Status verified 2023-10

CONDITIONS: Laryngotracheal Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Laryngotracheal Stenosis: Patients with laryngotracheal stenosis will have pressure sensors placed proximal and distal to the stenosis. Pressure and air flow will be measured
  Interventions: Diagnostic Test: Measure Airway Resistance Across Stenosis

INTERVENTIONS:
Diagnostic Test: Measure Airway Resistance Across Stenosis — Measure pressure and air flow Across Stenosis

SUMMARY:
This research is being done to determine the resistance across stenosis in the airway.

DETAILED DESCRIPTION:
There is significant utility in objectively measuring airflow as subjects, undergoing endoscopic laryngeal surgery, commonly have difficulties with airflow secondary to their stenosis. Easier and quicker quantification will tailor diagnosis and treatment. In order to obtain an objective measure of airflow in these participants, we will place a 20-gauge angiocatheter needle into the airway. The catheter will be in situ for a short duration during several spontaneous and non-spontaneous breaths. This will be achieved via the existing tracheostomy stoma or percutaneously via the cricothyroid membrane. This technique is commonly used to access the muscles of the larynx, however, the primary purpose will be to measure airflow in this setting.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years or older that require outpatient endoscopic laryngeal airway surgery, in the operating room, at a tertiary academic center.

Exclusion Criteria:

* Pregnancy (status will be determined by a urine test as part of standard clinical care in the preoperative setting)
* Patients that are not cleared for surgery by the preoperative evaluation
* Patients with severe laryngotracheal stenosis
* Patients who are morbidly obese (BMI > 40)
* Patients with lung disease (asthma, COPD)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients that require outpatient endoscopic laryngeal airway surgery in the operating room.
Sampling Method: Non-Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2017-03-29 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-05-31 (Actual)

PRIMARY OUTCOMES:
Pressure (cm H20) | Up to One Year
  Using a pressure gauge to measure pressure at locations in the airway

SECONDARY OUTCOMES:
Flow Rate (L/min) | Up to One Year
  using a flow sensor to measure low rate at locations in airway

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Hillel, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States